CLINICAL TRIAL: NCT00503750
Title: Phase II Neoadjuvant Trial of Trastuzumab in Combination With Dose-Dense ABI-007 (Abraxane™) Followed by Vinorelbine for HER2 Overexpressing Early Stage Breast Cancer
Brief Title: Phase II Neoadjuvant Trial of Trastuzumab in Combination With Dose-Dense ABI-007 (Abraxane™)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Ruth O'Regan, Principal Investigator, Emory University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0495-2006
Record Dates: First submitted 2007-07-17; First posted 2007-07-19 (Estimated); Results first posted 2012-06-14 (Estimated); Last update posted 2012-06-25 (Estimated); Status verified 2012-06

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Albumin-Bound Paclitaxel; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Trastuzumab and Abraxane followed Trastuzumab and Vinorelbine (Active Comparator): Patients will be treated sequentially with preoperative trastuzumab and dose-dense ABI-007 followed by trastuzumab in combination with vinorelbine. Trastuzumab will be administered as a one-time loading dose of 4 mg/kg as a 90 minute infusion, followed by 20 weekly treatments at 2 mg/kg as a 30 minute infusion. ABI-007 will be administered every 2 weeks at a dose of 260mg/m2 as 30 minute infusion on the same days as trastuzumab for a total of 4 cycles (weeks 1 -8). Growth factor support with pegfilgrastim (Neulasta®) is required 24 to 48 hours following completion of each cycle of ABI-007. Beginning week 9, patients will then receive weekly vinorelbine at a dose of 25mg/m2 for 12 weeks on the same day as trastuzumab for a total of 4 cycles (weeks 9-20). As per standard treatment of HER2-positive breast cancers, patients will continue to receive trastuzumab every 3 weeks at 6 mg/kg beginning week 21 through week 52.
  Interventions: Drug: Pre operativeTrastuzumab; Drug: ABI-007 (Abraxane); Drug: Vinorelbine

INTERVENTIONS:
Drug: Pre operativeTrastuzumab — Trastuzumab one-time loading dose of 4 mg/kg as 90 minute infusion, followed by 20 weekly treatments at 2 mg/kg as 30 minute infusion.
  As per standard treatment of HER2-positive breast cancers, patients will continue to receive trastuzumab every 3 weeks at 6 mg/kg beginning week 21 through week 52.
Drug: ABI-007 (Abraxane) — ABI-007 will be administered every 2 weeks at a dose of 260mg/m2 as 30 minute infusion on the same days as trastuzumab for a total of 4 cycles (weeks 1 -8).
Drug: Vinorelbine — Beginning week 9, patients will then receive weekly vinorelbine at a dose of 25mg/m2 for 12 weeks on the same day as trastuzumab for a total of 4 cycles (weeks 9-20).

SUMMARY:
This is a phase II one arm study. Patients with HER2 (Human Epidermal Growth Factor Receptor 2)positive early stage breast cancer will receive ABI-007 and vinorelbine in combination with trastuzumab before having breast surgery.

DETAILED DESCRIPTION:
This is a phase II one arm study. Patients with HER2(Human Epidermal Growth Factor Receptor 2) positive early stage breast cancer will receive ABI-007 and vinorelbine in combination with trastuzumab before having breast surgery.

Approximately 50 patients will take part at multi-sites with potentially 20 patients participating at the Emory Winship Cancer Institute, Grady Memorial Hospital, and Emory Crawford Long Hospital in Atlanta, Georgia.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed invasive breast carcinoma.
* Early stage breast cancer - stage I (tumor size greater than 1 cm), II and IIA.
* 3+ HER2 overexpression by IHC or 2+ HER2 overexpression and FISH positivity.
* Patients must have measurable disease as defined by palpable lesion with both diameters greater than or equal to 1 cm measurable with caliper and/or a positive mammogram or ultrasound with at least one dimension greater than or equal to 1 cm. Bilateral mammogram and clip placement is required for study entry. Baseline measurements of the indicator lesions must be recorded on the patient registration form. To be valid for baseline, the measurements must have been made within the 14 days (4-6 weeks for x-rays and scans) immediately preceding patient's entry in study.
* ECOG performance status 0 to 2 within 14 days of study entry.
* Normal (greater than 50%) left ventricular ejection fraction (LVEF) by MUGA scan or echocardiography.
* Must be 18 years of age or older.
* Women or men of childbearing potential must use a reliable and appropriate contraceptive method. Postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential.
* Final eligibility for a clinical trial is determined by the health professionals conducting the trial.

Exclusion Criteria:

* Evidence of disease outside the breast or chest wall, except ipsilateral axillary lymph nodes.
* Prior chemotherapy, hormonal therapy, biologic therapy or radiation therapy for breast cancer. Patients with history of DCIS are eligible if they were treated with surgery alone.
* Medical, psychological, or surgical condition which the investigator feels might compromise study participation.
* Pregnant or lactating women are not eligible.
* Patients with history of previous or current malignancy at other sites with the exception of adequately treated carcinoma in situ of the cervix or basal or squamous cell carcinoma of the skin. Patients with a history of other malignancies who remain disease free for greater than five years are eligible.
* Evidence of sensory and/or peripheral neuropathy.
* Serious, uncontrolled, concurrent infections.
* Major surgery within 4 weeks of the start of study treatment without complete recovery.
* Final eligibility for a clinical trial is determined by the health professionals conducting the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2008-04; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruth O'Regan, MD, Principal Investigator — Emory University Winship Cancer Institute
Locations (2):
- United States (2):
  - Piedmont Hospital Research Institute, Atlanta, Georgia
  - Emory University Winship Cancer Institute, Atlanta, Georgia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Trastuzumab and Abraxane Followed Trastuzumab and Vinorelbine
Started | 27
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Trastuzumab and Abraxane Followed Trastuzumab and Vinorelbine
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 0
Age Continuous [Median (Full Range); unit: years] | 49 [34 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Pathologic Response.
Description: Pathologic complete response (pCR): Absence of invasive breast cancer in the breast (mastectomy or lumpectomy) specimen at the time of definitive surgery. Presence of in situ cancer alone will be considered a pCR.
  Although clinical examination is the primary method of determining response, radiologic assessments (mammogram, ultrasound ± MRI) may be used to confirm response/non-response.
Time Frame: assess at 8 weeks
Measure: Number; unit: participants
Arm/Group | Trastuzumab and Abraxane Followed Trastuzumab and Vinorelbine
Number analyzed (Participants) | 27
participants | 13

2. Secondary Outcome: Number of Participants Who Had Complete Clinical Resposnse, Partial Response and Stable Disease.
Description: Complete clinical response (CCR): complete disappearance of all measurable malignant disease. No new malignant lesion, disease-related symptoms or evidence of non-evaluable disease.
  Partial response (PR): Reduction by at least 50% of the sum of the products of the longest perpendicular diameters of all measurable lesions.
  Stable disease (SD): For bidimensionally measurable disease, no decrease or <25% increase in the sum of the products of the longest perpendicular diameters of all measurable lesions.
Time Frame: clinic examination every 2 weeks, evaluated every 3 months for 2 years post-op
Measure: Number; unit: participants
Arm/Group | Trastuzumab and Abraxane Followed Trastuzumab and Vinorelbine
Number analyzed (Participants) | 27
participants
  Complete Response | 20
  Partial Response | 7
  Stable Disease | 0

ADVERSE EVENTS:
Arm/Group | Trastuzumab and Abraxane Followed Trastuzumab and Vinorelbine
Serious Adverse Events (participants affected / at risk) | 12/27
Other Adverse Events (participants affected / at risk) | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab and Abraxane Followed Trastuzumab and Vinorelbine (N=27)
Neuropathy (Nervous system disorders) | 3
Neutropenia (Nervous system disorders) | 6
Febrile Neutropenia (Nervous system disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Fatigue (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab and Abraxane Followed Trastuzumab and Vinorelbine (N=27)
Neuropathy (Blood and lymphatic system disorders) | 20
Neutropenia (Nervous system disorders) | 4
Febrile Neutropenia (Blood and lymphatic system disorders) | 0
Fatigue (General disorders) | 18
Nausea (Gastrointestinal disorders) | 11
Myalgias/Arthralgias (Musculoskeletal and connective tissue disorders) | 20
Liver Tests (Hepatobiliary disorders) | 12
Nail changes (Skin and subcutaneous tissue disorders) | 3
Anemia (Blood and lymphatic system disorders) | 14
Stomatitis (General disorders) | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Diarrhea (Gastrointestinal disorders) | 7
Constipation (Gastrointestinal disorders) | 9
Headache (General disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes